CLINICAL TRIAL: NCT01056107
Title: Effect of ROSE-010 on Gastrointestinal Motor Functions in Female Patients With Constipation Predominant Irritable Bowel Syndrome (C-IBS)
Brief Title: Effects of ROSE-010 on GI Transit in Constipation Predominant Irritable Bowel Syndrome (C-IBS) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Rose Pharma A/S (Unknown); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-005871; UL1RR024150 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Irritable Bowel Syndrome Constipation Predominant
Keywords: Constipation, Irritable Bowel Syndrome (IBS), Glucagon Like Peptide analogue
MeSH Terms: conditions — Constipation; Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens | interventions — glucagon-like peptide (7-37), valyl(10)-; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ROSE-010 30 mcg (Experimental): A glucagon-like peptide-1 (GLP-1) analogue. Subjects received a ROSE-010 30 mcg subcutaneous injection daily for 3 consecutive days and on 1 day 2-10 days later.
  Interventions: Drug: ROSE-010
- ROSE-010 100 mcg (Experimental): A glucagon-like peptide-1 (GLP-1) analogue. Subjects received a ROSE-010 100 mcg subcutaneous injection daily for 3 consecutive days and on 1 day 2-10 days later.
  Interventions: Drug: ROSE-010
- ROSE-010 300 mcg (Experimental): A glucagon-like peptide-1 (GLP-1) analogue. A glucagon-like peptide-1 (GLP-1) analogue. Subjects received a ROSE-010 300 mcg subcutaneous injection daily for 3 consecutive days and on 1 day 2-10 days later.
  Interventions: Drug: ROSE-010
- Placebo (Placebo Comparator): Subjects received a matching placebo subcutaneous injection daily for 3 consecutive days and on 1 day 2-10 days later.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ROSE-010 — The study medication was used in 30 mcg, 100 mcg, and 300 mcg subcutaneous injections daily, depending upon study arm.
  Other Names: Glucagon-like peptide-1 (GLP-1) analogue
  Arms: ROSE-010 100 mcg; ROSE-010 30 mcg; ROSE-010 300 mcg
Drug: Placebo — Placebo subcutaneous injection daily
  Other Names: Glucagon-like peptide-1 (GLP-1) analogue
  Arms: Placebo

SUMMARY:
This trial will study the effects of an investigational (not FDA approved) medication, ROSE-010, on the movement of food through the stomach, small intestine and colon in females with constipation predominant irritable bowel syndrome (C-IBS).

The study hypothesis is that ROSE-010 will delay gastric emptying of solids and enhances gastric accommodation without retarding colonic transit in female patients with C-IBS.

DETAILED DESCRIPTION:
Methodology

Female patients with C-IBS will be screened for eligibility and informed about the study at the initial screening visit Visit 1. Within two weeks of Visit 1, eligible patients will be randomized to study medication, either 30 mcg, 100 mcg or 300 mcg ROSE-010 or placebo administered via abdominal subcutaneous (s.c.) injection for a total of four days, three consecutive days during transit scintigraphy and once prior to SPECT imaging. The allocation to treatment group will be concealed.

Study medication will be administered at Visits 2, 3, and 4, the days of scintigraphic assessment of gastric, small bowel and colonic transit of solids performed over a 48 hour period.

Within two to seven days of Visit 4, patients will be instructed to return for administration of a final injection of study medication followed by SPECT gastric accommodation measurements (Visit 5). Within seven to ten days of Visit 5, patients will return for Visit 6, final safety monitoring and an exit interview with study staff.

Investigational product, dosage and mode of administration

Patients will receive placebo or 30 mcg, 100 mcg or 300 mcg ROSE-010 administered s.c. in the abdomen once on Visit 2, immediately before the standardized breakfast meal, fifteen minutes before the first camera image is obtained. Study medication will be administered fifteen minutes before camera images obtained on Visits 3 and 4. Study medication will be administered immediately after the first fasting scan is obtained and before the second fasting scan during SPECT at Visit 5.

Duration of treatment

ROSE-010 or matching placebo will be administered via abdominal s.c injection once daily for three consecutive days and one final day two to seven days later, over a ten-day interval.

Duration of patients involvement in the study

Each patient will attend six visits at the clinic during a period of two to four weeks.

Efficacy assessments

1. Scintigraphic gastrointestinal and colonic transit
2. Technetium-99m (99mTc) SPECT measurement of gastric volumes
3. Assessment of stool frequency and consistency made by the patient using the Bowel Pattern Diary

Safety assessments

The following safety assessments will be performed:

1. Laboratory safety tests, including a complete blood count (CBC), a comprehensive metabolic panel (CMP), and urinalysis (UA) at Visit 1 (study entry) and Visit 6 (study exit)
2. A physical examination by a study physician at Visit 1
3. Weight and vital signs (including temperature, pulse, blood pressure and respiration rate) at every visit
4. Urine pregnancy tests performed at Visit 1 and within 48 hours prior to receipt of radiation at Visit 2 transit test and Visit 5 SPECT test
5. Interview for concomitant medications and adverse events at every visit

Statistical methods

An analysis of covariance (ANCOVA) will be used to compare transit parameters and gastric volumes among the treatment groups. If necessary a suitable transformation for potential skewness in the distributions of measured volumes may be used (e.g., ANCOVA on ranks or log volumes). If ANCOVA shows a p value less than or equal to 0.10, then both the 100 mcg and 300 mcg doses will be compared to placebo (p value less than or equal to 0.25). Dunnett's Test will be used to compare each dose group with placebo. Since each of the primary endpoints assesses a separate hypothesis regarding the effects of ROSE-010, no adjustment in the alpha level for testing multiple types of endpoints is anticipated, and a two-sided significance level of 0.05 will be used in each ANCOVA model.

Analysis data sets

The primary analyses will follow the intent to treat (ITT) paradigm with all patients randomized included in the analyses. Those patients with missing response values will have their missing values imputed via the overall (patients with non-missing data) mean and a corresponding adjustment in the ANCOVA residual error variance degrees of freedom (subtracting one for each missing value imputed). Safety data will be presented for all patients receiving investigational product.

ELIGIBILITY:
Inclusion criteria:

1. Female aged 18-65 years old inclusive.
2. A previous diagnosis of IBS according to Rome III criteria to include those patients who have had recurrent abdominal pain or discomfort for the at least the six months prior to diagnosis and currently at least three days per month in the last three months associated with two or more of the following:

   1. improvement with defecation
   2. onset associated with a change in the frequency of stool
   3. onset associated with a change in form (appearance) of stool.
3. Constipation predominant type IBS as defined by one or more of the following:

   1. fewer than three spontaneous complete bowel movements per week
   2. hard or lumpy stools more than 25% of the time
   3. straining during a bowel movement more than 25% of the time.
4. A normal rectal exam result on file within the past two years or performed at screen to exclude the possibility of an evacuation disorder. Examination must exclude findings suggestive of an evacuation disorder such as high sphincter tone at rest, failure of perineal descent by more than one centimeter on straining and last, spasm, tenderness or paradoxical contraction of the puborectalis muscles.
5. Females of child bearing potential (those who have not experienced a bilateral tubal ligation, hysterectomy or menopause) must use an acceptable method of contraception during the study. Acceptable methods are surgical sterilization, hormonal methods such as oral contraceptives, Norplant and Depo-Provera, double barrier method such as a condom and spermicide, and an intrauterine device (IUD). Abstinent females may participate if they agree to use the double barrier method should they become sexually active during the study.
6. Able to provide written informed consent prior to any study procedures being performed.

Exclusion Criteria:

1. Female patients who are pregnant or breast-feeding.
2. Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders other than C-IBS.
3. Unable to withdraw medications 48 hours prior to the study: any medication that alters GI transit including but not limited to laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants and serotonin-norepinephrine reuptake inhibitors (SNRIs); analgesic drugs including opiates, nonsteroidal anti-inflammatory drugs (NSAIDs), and COX 2 inhibitors (Note: Tylenol is permitted), GABAergic agents and benzodiazepines. Note: All other concomitant medications will be reviewed on a case by case basis by the study physicians.
4. Clinical evidence (including but not limited to a clinically significant abnormal physical exam, ECG or laboratory result in the past medical record) or current clinically significant abnormal physical exam or laboratory test result that could indicate significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other diseases that interfere with the objectives of the study. If a laboratory test result is abnormal and clinically significant, it may be repeated once at the discretion of the PI. If the laboratory test result remains abnormal and clinically significant, the patient will be referred to a primary care physician for further evaluation.
5. Patients who are considered by the Investigator to be alcoholics not in remission or known substance abusers.
6. Patients who have participated in another clinical study within the past 30 days.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Camilleri M, Vazquez-Roque M, Iturrino J, Boldingh A, Burton D, McKinzie S, Wong BS, Rao AS, Kenny E, Mansson M, Zinsmeister AR. Effect of a glucagon-like peptide 1 analog, ROSE-010, on GI motor functions in female patients with constipation-predominant irritable bowel syndrome. Am J Physiol Gastrointest Liver Physiol. 2012 Jul;303(1):G120-8. doi: 10.1152/ajpgi.00076.2012. Epub 2012 Apr 19. PMID 22517769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 52 subjects were enrolled, but 6 subjects were excluded because they did not meet eligibility criteria.
Groups:
- ROSE-010 300 Mcg: A glucagon-like peptide-1 (GLP-1) analogue. Subjects received a ROSE-010 300 mcg subcutaneous injection daily for 3 consecutive days and on 1 day 2-10 days later.
Period: Overall Study
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Started | 11 | 11 | 12 | 12
Completed | 11 | 10 | 9 | 12
Not Completed | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 43.4 (6.0) | 40.2 (11.7) | 42.0 (11.9) | 43.8 (8.0) | 42.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 12 | 12 | 46
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 12 | 12 | 46
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (3.8) | 26.4 (5.5) | 26.4 (4.8) | 27.7 (4.0) | 26.9 (4.5)
Stool frequency [Mean (Standard Deviation); unit: Stools/day] | 0.7 (0.3) | 1.0 (0.8) | 0.8 (0.6) | 0.7 (0.4) | 0.8 (0.5)
Stool Consistency [Mean (Standard Deviation); unit: units on a scale] — The subjects rated their stool consistency using the Bristol Stool Scale. The Bristol Stool Scale is a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea.
  units on a scale | 2.8 (1.1) | 3.0 (0.8) | 2.8 (1.8) | 2.4 (0.9) | 2.7 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Colonic Transit, Colonic Geometric Center at 24 Hours
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
Time Frame: 24 hours (Visit 3 = Day 1)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
units on a scale | 2.39 (0.22) | 2.37 (0.41) | 2.02 (0.23) | 1.76 (0.14)

2. Primary Outcome: Change Between Postprandial and Fasting Whole Gastric Volume by Technetium-99m (99mTc)-SPECT Imaging (Gastric Accommodation)
Description: A noninvasive SPECT method was used to measure gastric volume during fasting and 32 min after a liquid nutritional supplement meal. Subjects reported to the clinic after an overnight fast. 99mTC was giving by an intravenous injection in the forearm. The first fasting scan was obtained, and the study medication was given s.c. After 10 min, a 2nd fasting post medication scan was obtained, and the meal consumed; then two serial postprandial scans were obtained. Each scan required 9-12 min. Tomographic images of the gastric wall were obtained throughout the long axis of the stomach using a dual-head gamma camera that rotates around the body. This allows assessment of the radiolabeled circumference of the gastric wall, rather than the intragastric content. For this outcome measure, the scans for the "fasting volume" and 2 "postprandial volumes" were used. The 2 postprandial (PP) volumes were averaged. Change was calculated as (PP - Fasting = gastric accommodation).
Time Frame: approximately 1 hour after 99mTC injection, approximately 30 min after liquid meal (Visit 5 = approximately 2-10 days after Visit 4)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: mL
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
mL | 532.2 (36.6) | 575.6 (19.4) | 515.2 (52.5) | 532.8 (22.8)

3. Primary Outcome: Half Time (t1/2) of Gastric Emptying of Solids Measured by Scintigraphy (Gastric Transit)
Description: Half time (t1/2) of gastric emptying (GE) of solids is the time for half of the ingested solids or liquids to leave the stomach. The scintigraphy for GE t1/2 was done on Visit 2 (Day 0 of the study), the first day of scintigraphy.
Time Frame: approximately 2 hours after radiolabeled meal is ingested (Visit 2 = Day 0)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: minutes
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
minutes | 151.8 (10.4) | 172.6 (7.1) | 210.7 (8.6) | 136.9 (7.2)
Statistical Analysis 1: Comparison: ROSE-010 100 Mcg vs Placebo; Test type: Superiority or Other; p = 0.0075, Dunnett's test
Statistical Analysis 2: Comparison: ROSE-010 300 Mcg vs Placebo; Test type: Superiority or Other; p < 0.001, Dunnett's test

4. Secondary Outcome: Gastric Residual at 2 and 4 Hours Measured by Scintigraphy
Description: The gastric residual will be calculated as the proportion of isotope remaining in the stomach (at 2 and 4 hours).
Time Frame: 2 hours, 4 hours (Visit 2 = Day 0)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: proportion of isotope in the stomach
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
proportion of isotope in the stomach
  Gastric residual at 2 hours | 0.66 (0.42) | 0.76 (0.03) | 0.86 (0.03) | 0.59 (0.04)
  Gastric residual at 4 hours | 0.14 (0.03) | 0.16 (0.03) | 0.30 (0.06) | 0.12 (0.03)

5. Secondary Outcome: Colonic Geometric Center at 4 h Measured by Scintigraphy
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool. (Note: when there is no radio isotope in the colon (e.g., at 4 hours) the geometric center values are recorded as "zero," thus the mean values can be less than one.)
Time Frame: 4 hours (Visit 2 = Day 0)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
units on a scale | 0.70 (0.20) | 0.47 (0.16) | 0.57 (0.17) | 0.53 (0.17)

6. Secondary Outcome: Colonic Filling at 6 h Measured by Scintigraphy
Description: Percent of the radio-labeled meal that reached the colon at 6 hours, indirectly reflecting small bowel transit time.
Time Frame: 6 hours (Visit 2 = Day 0)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: percentage of meal
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
percentage of meal | 47.6 (7.4) | 54.4 (7.8) | 48.0 (10.0) | 53.5 (4.8)

7. Secondary Outcome: Ascending Colon Emptying Half-time (AC t1/2) Measured by Scintigraphy
Description: Ascending colon emptying half-time will be estimated by power exponential analysis of the proportionate emptying over time of counts from the colon. The primary data for this analysis will be the proportion of decay and depth-corrected counts in the ascending colon on the hourly scans on the first day of transit measurement and the 48 hour data.
Time Frame: 48 hours (Visit 4 = Day 2)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: hours
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
hours | 14.5 (1.6) | 14.8 (3.7) | 17.1 (4.0) | 19.3 (3.2)

8. Secondary Outcome: Colonic Transit, Colonic Geometric Center at 48 h Measured by Scintigraphy, as Compared to Placebo.
Description: as for outcome 1
Time Frame: 48 hours (Visit 4 = Day 2)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
units on a scale | 3.69 (0.23) | 3.79 (0.33) | 3.36 (0.37) | 2.67 (0.26)

9. Secondary Outcome: Stool Frequency
Description: Stool frequency was self reported in a Bowel Pattern Diary. The bowel pattern diary was dispensed at the screening visit, and the completed bowel pattern diary was collected at the completion of the study.
Time Frame: screening visit (Visit 1), 34 days (Visit 6)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: Stools/day
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
Stools/day | 0.75 (0.09) | 1.13 (0.17) | 0.88 (0.15) | 0.70 (0.05)

10. Secondary Outcome: Stool Consistency Post Treatment
Description: The subjects rated their stool consistency using the 7-point Bristol Stool Scale. The Bristol Stool Scale is a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea. The Bristol stool form was part of the bowel pattern diary, which was dispensed at the screening visit, and the completed bowel pattern diary was collected at the completion of the study.
Time Frame: 34 days (Visit 6)
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Number analyzed (Participants) | 11 | 11 | 12 | 12
units on a scale | 2.93 (0.33) | 2.96 (0.36) | 2.93 (0.47) | 3.05 (0.32)

ADVERSE EVENTS:
Time Frame: Subjects were assessed for adverse events at every study visit, approximately over 22 days.
Arm/Group | ROSE-010 30 Mcg | ROSE-010 100 Mcg | ROSE-010 300 Mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/11 | 10/11 | 11/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ROSE-010 30 Mcg (N=11) | ROSE-010 100 Mcg (N=11) | ROSE-010 300 Mcg (N=12) | Placebo (N=12)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (8) | 9 (9) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Dry heaving (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal cramp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 3 (3) | 4 (4) | 2 (2)
Drowsiness (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Injection site rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No